CLINICAL TRIAL: NCT00271817
Title: Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin and Niacin (Extended Release Tablet) Co-Administered in Patients With Type IIa or Type IIb Hyperlipidemia
Brief Title: To Evaluate Ezetimibe/Simvastatin and Niacin (Extended Release Tablet) in Patients With Type IIa or Type IIb Hyperlipidemia (0653A-091)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-091; 2005_091
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin; Niacin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part 1 - Arm 1 (Active Comparator): ezetimibe/simvastatin combination tablet + niacin (ER)
  Interventions: Drug: Comparator: ezetimibe/simvastatin + niacin (ER)
- Part 1 -Arm 2 (Active Comparator): ezetimibe/simvastatin
  Interventions: Drug: Comparator: ezetimibe (+) simvastatin; Drug: Comparator: Placebo to Niacin (ER)
- Part 1 - Arm 3 (Active Comparator): Niacin (ER)
  Interventions: Drug: Comparator: Placebo to ezetimibe/simvastatin; Drug: Comparator: niacin (ER) tablet
- Part 2 - Arm 1 (Active Comparator): ezetimibe/simvastatin combination tablet + niacin (ER)
  Interventions: Drug: Comparator: ezetimibe/simvastatin and niacin (ER)
- Part 2 - Arm 2 (Placebo Comparator): ezetimibe/simvastatin combination tablet + niacin (Pbo)
  Interventions: Drug: Comparator: ezetimibe and simvastatin; Drug: Comparator: Placebo to niacin (ER)

INTERVENTIONS:
Drug: Comparator: ezetimibe/simvastatin + niacin (ER) — ezetimibe/simvastatin 10/20mg tablet + niacin (ER) tablet, titrating to 2g, po qd. Treatment time will be ~24 weeks
  Arms: Part 1 - Arm 1
Drug: Comparator: Placebo to ezetimibe/simvastatin — ezetimibe/simvastatin (Pbo) tablet. Treatment time will be ~24 weeks.
  Arms: Part 1 - Arm 3
Drug: Comparator: niacin (ER) tablet — niacin (ER) tablet, titrating to 2g, po qd. Treatment time will be ~24 weeks
  Arms: Part 1 - Arm 3
Drug: Comparator: ezetimibe (+) simvastatin — ezetimibe/simvastatin 10/20mg tablet. Treatment time will be ~24 weeks.
  Arms: Part 1 -Arm 2
Drug: Comparator: Placebo to Niacin (ER) — Niacin (ER) (Pbo) tablet. Treatment time will be ~24 weeks.
  Arms: Part 1 -Arm 2
Drug: Comparator: ezetimibe/simvastatin and niacin (ER) — ezetimibe/simvastatin 10/20mg tablet + niacin (ER) tablet 2g, po qd. Treatment time will be ~40 additional weeks for a total of 64 weeks
  Arms: Part 2 - Arm 1
Drug: Comparator: ezetimibe and simvastatin — ezetimibe/simvastatin 10/20mg tablet. Treatment time will be ~40 additional weeks for a total of 64 weeks
  Arms: Part 2 - Arm 2
Drug: Comparator: Placebo to niacin (ER) — Niacin (ER) (Pbo) tablet. Treatment time will be ~40 additional weeks for a total of 64 weeks
  Arms: Part 2 - Arm 2

SUMMARY:
To evaluate the efficacy and safety of ezetimibe/simvastatin and niacin in patients with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Patient with LDL-C of 130 through 190 mg/dL and Triglycerides less than or equal to 500 mg/dL
* Patient willing to be on a low-cholesterol diet

Exclusion Criteria:

* Pregnant or lactating women or intending to become pregnant
* Patient with sensitivity or intolerance to ezetimibe, simvastatin, or ezetimibe/simvastatin combination tablet
* Patient with sensitivity or intolerance ro niacin, any component or niacin extended release or aspirin
* Patient for whom discontinuation of existing lipid-lowering therapy treatment poses an unacceptable risk

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guyton JR, Brown BG, Fazio S, Polis A, Tomassini JE, Tershakovec AM. Lipid-altering efficacy and safety of ezetimibe/simvastatin coadministered with extended-release niacin in patients with type IIa or type IIb hyperlipidemia. J Am Coll Cardiol. 2008 Apr 22;51(16):1564-72. doi: 10.1016/j.jacc.2008.03.003. PMID 18420099
- [Derived] Le NA, Jin R, Tomassini JE, Tershakovec AM, Neff DR, Wilson PW. Changes in lipoprotein particle number with ezetimibe/simvastatin coadministered with extended-release niacin in hyperlipidemic patients. J Am Heart Assoc. 2013 Aug 7;2(4):e000037. doi: 10.1161/JAHA.113.000037. PMID 23926117
- [Derived] Guyton JR, Fazio S, Adewale AJ, Jensen E, Tomassini JE, Shah A, Tershakovec AM. Effect of extended-release niacin on new-onset diabetes among hyperlipidemic patients treated with ezetimibe/simvastatin in a randomized controlled trial. Diabetes Care. 2012 Apr;35(4):857-60. doi: 10.2337/dc11-1369. Epub 2012 Feb 14. PMID 22338103

RESULTS

PARTICIPANT FLOW:
Groups:
- Niacin: (Part 1): Niacin titrated to 2000 mg taken orally once daily for 24 weeks. During the first 12 weeks of the study, patients randomized to the niacin containing arms started taking niacin 500 mg and had their niacin dose increased 500 mg every 4 weeks to 2000 mg. Patients in this treatment group were ramdomly reassigned for Part 2 of the study to one of two treatment groups- two-thirds of the patients enrolled in the niacin treatment group were randomly assigned to receive ezetimibe/simvastatin + niacin (ER) and the other one-third were randomly assigned to receive ezetimibe/simvastatin alone.
- Ezetimibe/Simvastatin: (Part 1): Ezetimibe/Simvastatin 10/20 mg taken orally once daily for 24 weeks.
  (Part 2): Ezetimibe/Simvastatin 10/20 mg taken orally once daily for 40 additional weeks for a total of 64 weeks.
- Ezetimibe/Simvastatin + Niacin: (Part 1): Ezetimibe/Simvastatin 10/20 mg + Niacin (titrated to 2000 mg as noted above) taken orally once daily for 24 weeks.
  (Part 2): Ezetimibe/Simvastatin 10/20 mg + Niacin 2000 mg taken orally once daily for 40 additional weeks for a total of 64 weeks.
Period: Part 1
Arm/Group | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Started | 272 | 272 | 676
Completed | 166 (6 patients who completed Part 1 did not continue to Part 2; 1 patient never received drug in Part 2) | 213 (1 patient who completed Part 1 did not continue to Part 2) | 391 (11 patients who completed Part 1 did not continue to Part 2)
Not Completed | 106 | 59 | 285
Not completed — Adverse Event | 68 | 25 | 156
Not completed — Lost to Follow-up | 6 | 8 | 24
Not completed — Protocol Violation | 5 | 4 | 7
Not completed — Patient Moved | 3 | 1 | 5
Not completed — Withdrawal by Subject | 23 | 17 | 45
Not completed — LDL < 50 mg/dL | 1 | 4 | 48
Period: Part 2
Arm/Group | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Started | 0 (Patients completing the niacin group in Part 1, were re-allocated to one of the two arms in Part 2) | 266 (Includes 54 patients re-allocated from the niacin group in Part 1) | 485 (Includes 105 patients re-allocated from the niacin group in Part 1)
Completed | 0 | 234 | 401
Not Completed | 0 | 32 | 84
Not completed — Adverse Event | 0 | 17 | 33
Not completed — Lack of Efficacy | 0 | 1 | 6
Not completed — Lost to Follow-up | 0 | 6 | 18
Not completed — Protocol Violation | 0 | 3 | 5
Not completed — Patient Moved | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 13
Not completed — LDL < 50 mg/dL | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Niacin: (Part 1): Niacin titrated to 2000 mg taken orally once daily for 24 weeks. During the first 12 weeks of the study, patients randomized to the niacin containing arms started taking niacin 500 mg and had their niacin dose increased 500 mg every 4 weeks to 2000 mg.
- Total: Total of all reporting groups
Arm/Group | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin | Total
Number analyzed (Participants) | 272 | 272 | 676 | 1220
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.6) | 57.5 (10.3) | 56.9 (10.9) | 56.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 120 | 352 | 608
  Male | 136 | 152 | 324 | 612
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 11 | 4 | 11 | 26
  Black | 13 | 17 | 38 | 68
  Hispanic | 14 | 11 | 49 | 74
  Other | 3 | 0 | 2 | 5
  White | 231 | 240 | 576 | 1047
Body Mass Index [Number; unit: Participants]
  <25 kg/m2 | 48 | 39 | 135 | 222
  25 to <30 kg/m2 | 110 | 119 | 252 | 481
  30 to <40 kg/m2 | 97 | 94 | 251 | 442
  ≥ 40 kg/m2 | 16 | 19 | 34 | 69
  No BMI Data | 1 | 1 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to niacin extended release monotherapy on the percent change, from baseline in LDL-C after 24 weeks - 24 Week Measure Minus Baseline
Time Frame: Baseline and 24 Weeks
Population: The participant population for this analysis is the Completers Population. This includes all patients with a baseline value, who receive at least 24 weeks of active study therapy, and who have an on-treatment measurement at the maximum titrated dose per the protocol.
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Niacin: Niacin titrated to 2000 mg taken orally once daily for 24 weeks. During the first 12 weeks of the study, patients randomized to the niacin containing arms had their niacin titrated (increased 500 mg every 4 weeks to 2000 mg).
- Ezetimibe/Simvastatin + Niacin: Ezetimibe/Simvastatin 10/20 mg + Niacin (titrated to 2000 mg) taken orally once daily for 24 weeks.
Arm/Group | Niacin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 166 | 391
Percent change | -20.1 (1.3) | -58.5 (0.8)
Statistical Analysis 1: Comparison: Niacin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — A fixed sequence testing procedure was employed where testing followed a prespecified order and each subsequent hypothesis was tested at the 0.05 level of significance only if all previously tested hypotheses have been rejected; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -38.4, 95% CI [-41.4 to -35.4], Standard Error of Mean 1.5 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin

2. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to niacin extended release monotherapy on the percent change from baseline in non-HDL-C after 24 weeks - 24 week measure minus baseline
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Niacin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 166 | 391
Percent change | -22.0 (1.3) | -55.6 (0.8)
Statistical Analysis 1: Comparison: Niacin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -33.5, 95% CI [-36.5 to -30.6], Standard Error of Mean 1.5 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin

3. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein-Cholesterol (HDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in HDL-C after 24 weeks - 24 week measure minus baseline
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Ezetimibe/Simvastatin: Ezetimibe/Simvastatin 10/20 mg taken orally once daily for 24 weeks.
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 212 | 391
Percent change | 8.1 (1.3) | 30.2 (1.0)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = 22.1, 95% CI [18.8 to 25.3], Standard Error of Mean 1.6 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin

4. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in Triglycerides after 24 weeks - 24 week measure minus baseline
Time Frame: baseline and 24 Weeks
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 212 | 391
Percent change | 23.7 (29.7) | -42.5 (27.5)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment, baseline LDL-C, baseline TG and gender; Median Difference (Final Values) = -18.7, 95% CI [-22.6 to -14.7] — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin The median difference is based on the Hodges-Lehmann estimates of shift; The distribution-free 95% CI is based on Wilcoxon's rank sum test statistic

5. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein-Cholesterol (HDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in HDL-C after 64 weeks - 64 week measure minus baseline
Time Frame: Baseline and 64 weeks
Population: The analysis population is the modified intention-to-treat population, which includes patients that were randomized to ezetimibe/simvastatin + niacin or ezetimibe/simvastatin treatment groups and have a baseline measurement and at least on measurement beyond Week 24.
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Ezetimibe/Simvastatin: Ezetimibe/Simvastatin 10/20 mg taken orally once daily for 24 weeks. Ezetimibe/Simvastatin 10/20 mg taken orally once daily for 40 additional weeks for a total of 64 weeks.
- Ezetimibe/Simvastatin + Niacin: Ezetimibe/Simvastatin 10/20 mg + Niacin (titrated to 2000 mg) taken orally once daily for 24 weeks. Ezetimibe/Simvastatin 10/20 mg + Niacin 2000 mg taken orally once daily for 40 additional weeks for a total of 64 weeks.
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 207 | 369
Percent change | 9.0 (1.4) | 30.5 (1.1)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = 21.5, 95% CI [18.0 to 25.0], Standard Error of Mean 1.8 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin

6. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in Triglycerides after 64 weeks - 64 week measure minus baseline
Time Frame: Baseline and 64 weeks
Population: as for outcome 5
Measure: Median (Standard Deviation); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 207 | 369
Percent change | -26.8 (32.7) | -44.5 (26.9)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Median Difference (Final Values) = -17.6, 95% CI [-21.8 to -13.6] — Median difference = Ezetimibe/Simvastatin + Niacin minus Ezetimibe/Simvastatin The median difference is based on the Hodges-Lehmann estimates of shift; The distribution-free 95% CI is based on Wilcoxon's rank sum test statistic

7. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in non-HDL-C after 64 weeks - 64 week measure minus baseline
Time Frame: Baseline and 64 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 207 | 369
Percent change | -45.1 (1.3) | -52.4 (0.9)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -7.3, 95% CI [-10.4 to -4.2], Standard Error of Mean 1.6 — Median difference = Ezetimibe/Simvastatin + Niacin minus Ezetimibe/Simvastatin

8. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in LDL-C after 64 weeks - 64 week measure minus baseline
Time Frame: Baseline and 64 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 207 | 369
Percent change | -49.3 (1.3) | -54.0 (1.0)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -4.8, 95% CI [-8.0 to -1.5], Standard Error of Mean 1.6 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Ezetimibe/Simvastatin

9. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in LDL-C after 24 weeks - 24 week measure minus baseline
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 212 | 391
Percent change | -53.5 (1.2) | -58.5 (0.8)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -4.9, 95% CI [-7.7 to -2.1], Standard Error of Mean 1.4 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Niacin

10. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Ezetimibe/simvastatin co-administered with niacin extended release compared to ezetimibe/simvastatin monotherapy on the percent change from baseline in non-HDL-C after 24 weeks - 24 week measure minus baseline
Time Frame: Baseline and 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin
Number analyzed (Participants) | 212 | 391
Percent change | -47.9 (1.1) | -55.6 (0.8)
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Ezetimibe/Simvastatin + Niacin; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA with terms for treatment, baseline LDL-C, baseline TG, and gender; Mean Difference (Final Values) = -7.7, 95% CI [-10.4 to -5.0], Standard Error of Mean 1.4 — Mean difference = Ezetimibe/Simvastatin + Niacin minus Ezetimibe/Simvastatin

ADVERSE EVENTS:
Groups:
- Niacin: Niacin group from Part 1
- Ezetimibe/Simvastatin: Ezetimibe/Simvastatin group from Part 1
- Ezetimibe/Simvastatin + Niacin: Ezetimibe/Simvastatin + Niacin group from Part 1
- Ezetimibe/Simvastatin - Part 2: EZ/Simva group from Part 2 All-Treated Patient as Treated Population
- Ezetimibe/Simvastatin + Niacin - Part 2: Ezetimibe/Simvastatin + Niacin group from Part 2 All-Treated Patient as Treated Population
Arm/Group | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin | Ezetimibe/Simvastatin - Part 2 | Ezetimibe/Simvastatin + Niacin - Part 2
Serious Adverse Events (participants affected / at risk) | 8 | 13 | 16 | 29 | 59
Other Adverse Events (participants affected / at risk) | 121 | 428 | 185 | 175 | 505
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin | Ezetimibe/Simvastatin - Part 2 | Ezetimibe/Simvastatin + Niacin - Part 2
Anaemia (Blood and lymphatic system disorders) | 0/272 | 0/272 | 1/670 | 0/326 | 1/775
Aplastic Anaemia (Blood and lymphatic system disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Leukocytosis (Blood and lymphatic system disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Acute Coronary Syndrome (Cardiac disorders) | 0/272 | 1/272 | 1/670 | 1/326 | 1/775
Acute Myocardial Infarction (Cardiac disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Angina Pectoris (Cardiac disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Atrial Fibrillation (Cardiac disorders) | 0/272 | 1/272 | 0/670 | 0/326 | 1/775
Cardiac Failure Congestive (Cardiac disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Coronary Artery Disease (Cardiac disorders) | 0/272 | 0/272 | 1/670 | 1/326 | 2/775
Coronary Artery Stenosis (Cardiac disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Myocardial Infarction (Cardiac disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 1/775
Spondylolisthesis (Congenital, familial and genetic disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0/272 | 0/272 | 1/670 | 0/326 | 1/775
Pancreatic Mass (Gastrointestinal disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Pancreatitis (Gastrointestinal disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Chest Pain (General disorders) | 1/272 | 1/272 | 0/670 | 1/326 | 1/775
Non-Cardiac Chest Pain (General disorders) | 1/272 | 0/272 | 1/670 | 1/326 | 1/775
Pain (General disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Cholecystitis (Hepatobiliary disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Cholelithiasis (Hepatobiliary disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Anaphylactic Reaction (Immune system disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Abdominal Abscess (Infections and infestations) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Diverticulitis (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Herpes Zoster Oticus (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Influenza (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Osteomyelitis (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Perirectal Abscess (Infections and infestations) | 0/272 | 0/272 | 1/670 | 0/326 | 1/775
Pneumonia (Infections and infestations) | 1/272 | 0/272 | 0/670 | 0/326 | 1/775
Rocky Mountain Spotted Fever (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Sepsis (Infections and infestations) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Staphylococcal Infection (Infections and infestations) | 0/272 | 0/272 | 1/670 | 0/326 | 1/775
Viral Labyrinthitis (Infections and infestations) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Muscle Strain (Injury, poisoning and procedural complications) | 0/272 | 0/272 | 1/670 | 0/326 | 0/775
Ankle Fracture (Injury, poisoning and procedural complications) | 0/272 | 0/272 | 0/670 | 1/326 | 2/775
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Fibula Fracture (Injury, poisoning and procedural complications) | 0/272 | 1/272 | 0/670 | 1/326 | 1/775
Ligament Injury (Infections and infestations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Tibia Fracture (Injury, poisoning and procedural complications) | 0/272 | 1/272 | 0/670 | 1/326 | 1/775
Transaminases Abnormal (Investigations) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Dehydration (Metabolism and nutrition disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Hypovolaemia (Metabolism and nutrition disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/272 | 0/272 | 2/670 | 0/326 | 3/775
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/272 | 0/272 | 0/670 | 2/326 | 2/775
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 2/670 | 1/326 | 3/775
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/272 | 0/272 | 0/670 | 0/326 | 4/775
Cerebral Infarction (Nervous system disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Cerebrovascular Accident (Nervous system disorders) | 2/272 | 0/272 | 0/670 | 1/326 | 0/775
Cervical Cord Compression (Nervous system disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
Dizziness (Nervous system disorders) | 1/272 | 0/272 | 0/670 | 0/326 | 0/775
Paraesthesia (Nervous system disorders) | 0/272 | 0/272 | 1/670 | 0/326 | 1/775
Syncope (Nervous system disorders) | 0/272 | 0/272 | 2/670 | 0/326 | 3/775
Nephrolithiasis (Renal and urinary disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Renal Failure Acute (Renal and urinary disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Uterine Prolapse (Reproductive system and breast disorders) | 0/272 | 1/272 | 0/670 | 0/326 | 1/775
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/272 | 0/272 | 0/670 | 1/326 | 0/775
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0/272 | 1/272 | 0/670 | 1/326 | 0/775
Deep Vein Thrombosis (Vascular disorders) | 0/272 | 0/272 | 1/670 | 0/326 | 2/775
Thrombosis (Vascular disorders) | 0/272 | 0/272 | 0/670 | 0/326 | 1/775
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Niacin | Ezetimibe/Simvastatin | Ezetimibe/Simvastatin + Niacin | Ezetimibe/Simvastatin - Part 2 | Ezetimibe/Simvastatin + Niacin - Part 2
Constipation (Gastrointestinal disorders) | 0/272 | 0/670 | 0/272 | 8/326 | 10/775
Diarrhoea (Gastrointestinal disorders) | 9/272 | 27/670 | 10/272 | 12/326 | 47/775
Dyspepsia (Gastrointestinal disorders) | 0/272 | 0/670 | 0/272 | 7/326 | 7/775
Nausea (Gastrointestinal disorders) | 8/272 | 28/670 | 11/272 | 12/326 | 32/775
Vomiting (Gastrointestinal disorders) | 5/272 | 14/670 | 5/272 | 7/326 | 22/775
Fatigue (General disorders) | 7/272 | 13/670 | 6/272 | 9/326 | 18/775
Bronchitis (Infections and infestations) | 0/272 | 0/670 | 0/272 | 10/326 | 24/775
Gastroenteritis Viral (Infections and infestations) | 0/272 | 0/670 | 0/272 | 8/326 | 22/775
Nasopharyngitis (Infections and infestations) | 9/272 | 16/670 | 9/272 | 15/326 | 33/775
Sinusitis (Infections and infestations) | 7/272 | 21/670 | 5/272 | 17/326 | 35/775
Upper Respiratory Tract Infection (Infections and infestations) | 13/272 | 27/670 | 9/272 | 24/326 | 56/775
Urinary Tract Infection (Infections and infestations) | 7/272 | 6/670 | 3/272 | 8/326 | 10/775
Arthralgia (Musculoskeletal and connective tissue disorders) | 13/272 | 18/670 | 8/272 | 20/326 | 31/775
Back Pain (Musculoskeletal and connective tissue disorders) | 5/272 | 14/670 | 7/272 | 12/326 | 26/775
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8/272 | 10/670 | 7/272 | 11/326 | 16/775
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0/272 | 0/670 | 0/272 | 10/326 | 13/775
Myalgia (Musculoskeletal and connective tissue disorders) | 8/272 | 18/670 | 5/272 | 14/326 | 28/775
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7/272 | 16/670 | 8/272 | 12/326 | 25/775
Dizziness (Nervous system disorders) | 7/272 | 17/670 | 6/272 | 11/326 | 26/775
Headache (Nervous system disorders) | 8/272 | 13/670 | 12/272 | 14/326 | 18/775
Paraesthesia (Nervous system disorders) | 2/272 | 25/670 | 14/272 | 4/326 | 29/775
Insomnia (Psychiatric disorders) | 6/272 | 6/670 | 6/272 | 8/326 | 7/775
Cough (Respiratory, thoracic and mediastinal disorders) | 0/272 | 0/670 | 0/272 | 8/326 | 17/775
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3/272 | 8/670 | 6/272 | 7/326 | 12/775
Pruritus (Skin and subcutaneous tissue disorders) | 4/272 | 79/670 | 35/272 | 4/326 | 86/775
Rash (Skin and subcutaneous tissue disorders) | 4/272 | 32/670 | 15/272 | 6/326 | 41/775
Flushing (Vascular disorders) | 15/272 | 274/670 | 108/272 | 17/326 | 288/775
Hot Flush (Vascular disorders) | 3/272 | 15/670 | 5/272 | 4/326 | 18/775
Hypertension (Vascular disorders) | 0/272 | 0/670 | 0/272 | 9/326 | 3/775

LIMITATIONS AND CAVEATS:
Part 1 population is all patients enrolled in Part 1 of the study. Part 2 is those patients who received either niacin, ezetimibe/simvastatin, or ezetimibe/simvastatin + niacin during Part 1 until they finished the study at week 64 or discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.